CLINICAL TRIAL: NCT06909461
Title: The Effect of Pain Neuroscience Education on Physiotherapy Students' Knowledge, Attitudes and Behaviours Towards Pain: A Single-blinded Randomized Controlled Trial
Brief Title: The Effect of Pain Neuroscience Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Erhan Seçer, Principal Investigator, Celal Bayar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CBU-FTR-ES-05
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Student Education

STUDY DESIGN:
Intervention Model Description: A single-blinded randomized controlled trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Neuroscience Education Group (Active Comparator): The pain neuroscience education group will be receive a 70-min pain neuroscience education.
  Interventions: Other: Pain neuroscience education
- Control Group (Active Comparator): Red-flags education The control group will be receive a 70-min red-flags education.
  Interventions: Other: Red-flags education

INTERVENTIONS:
Other: Pain neuroscience education — The pain neuroscience education group will be receive a 70-min pain neuroscience education.
  Arms: Pain Neuroscience Education Group
Other: Red-flags education — The control group will be receive a 70-min red-flags education.
  Arms: Control Group

SUMMARY:
The aim of this study is to examine the effect of pain neuroscience education (PNE) on physiotherapy students' knowledge, attitudes and behaviors towards pain. A total of 52 physiotherapy students will be included in the study. Students will be randomly randomly assigned to either PNE group (n=26) or control group (CG) (n=26). The PNE group will be receive a 70-min PNE based on the explanations used in "Explain Pain". The CG group will be received an education about red-flags which are special screening questions for serious pathology. The red-flags education will be discussed tissue pathology and Waddell's triage for back pain classification.Neurophysiology and the biopsychosocial model will not be discussed. Before, immediately after, and 2-months after the education sessions all students will be completed four questionnaires, the Revised Neurophysiology Pain Questionnaire (RNP-Q), the Health Care Providers' Pain and Impairment Relationship Scale(HC-PAIRS), and the red-flags questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* volunteer to participate in study
* to studying in physiotherapy
* be able to read and understand Turkish

Exclusion Criteria:

- having received pain neuroscience education

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2025-04-05 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Pain neurophysiology knowledge | an hour
  The 12-item Revised Neurophysiology of Pain Questionnaire (RNP-Q) will be used to assess pain neurophysiology knowledge. Responses will be marked yes, no or undecided. One point is awarded for correct answers. Scores range from 0 to 12, with high scores indicating good knowledge. The RNPQ is a valid and reliable tool for assessing pain neurophysiology knowledge.

SECONDARY OUTCOMES:
Attitudes and behaviours | an hour
  The modified Health Care Providers' Pain and Impairment Relationship Scale (HC-PAIRS) will be used to assess students' attitudes and behaviours. This 13-item questionnaire uses a 7-point Likert scale (strongly disagree to strongly agree). Scores range from 13 to 91 with lower scores suggesting more positive attitudes. The HC-PAIRS has demonstrated good levels of validity and reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- Manisa Celal Bayar University, Manisa, Mani̇sa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided